CLINICAL TRIAL: NCT01667783
Title: Improving Diabetes Through Lifestyle and Surgery Study
Brief Title: Improving Diabetes Through Lifestyle and Surgery
Acronym: IDeaLS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK089557; R01DK089557 (NIH)
Record Dates: First submitted 2012-05-24; First posted 2012-08-17 (Estimated); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gastric Banding (Active Comparator): Laparoscopic Adjustable Gastric Banding
  Interventions: Procedure: Gastric Banding
- Medical Weight Loss (Active Comparator): Medical Weight Loss using a comprehensive lifestyle intervention consisting of diet (meal replacements), physical activity and behavioral techniques
  Interventions: Behavioral: Medical Weight Loss
- Gastric Bypass (Active Comparator): Roux-en-Y Gastric Bypass
  Interventions: Procedure: Gastric Bypass

INTERVENTIONS:
Procedure: Gastric Banding — Laparoscopic Adjustable Gastric Banding using the LapBand
  Arms: Gastric Banding
Behavioral: Medical Weight Loss — Weight loss intervention using diet (meal replacments), physical activity and behavioral techniques administered with weekly one-on-one counselling by dieticians
  Other Names: HMR meal replacements will be used
  Arms: Medical Weight Loss
Procedure: Gastric Bypass — Laparoscopic Roux-en-Y Gastric Bypass
  Arms: Gastric Bypass

SUMMARY:
Weight loss is effective in reducing many complications of obesity, with the majority of patients who undergo bariatric surgery having substantial improvements in their weight-related illnesses. The investigators propose a pilot study in 45 subjects with mild to moderate obesity to compare how losing 10% of initial body weight via one of three common weight loss strategies (medical weight loss with a low calorie diet, Roux-en-Y gastric bypass surgery, and adjustable gastric banding) affects diabetes. While the investigators do not expect this pilot study to provide definitive answers, it will provide valuable information to design a larger trial which will help guide therapy for people with mild-moderate obesity and substantial comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-40 kg/m2 at screening visit 1
* Age 21-64 years
* Insured by collaborating insurance plan (Employee Health Plan)
* Type 2 Diabetes
* Medically safe to undergo surgery and approved by a psychologist
* Able to exercise at a moderate level
* Able to give informed consent
* Willing to accept randomization to each group
* Able to communicate (both written and oral) in English
* Willing to use reliable method of birth control during study and ≥18 months postop (if applicable)

Exclusion Criteria:

* Prior bariatric surgery
* Prior gastric, small or large bowel, spleen, pancreas, kidney, or liver surgery, including large ventral hernia or previous large ventral hernia repair.
* Weight loss of ≥ 5% of body weight in the past 6 months
* Uncontrolled diabetes (HbA1c>8.5%)
* Untreated severe diabetic retinopathy
* Use of thiazolidinediones or insulin currently or within the past 3 months
* Uncontrolled blood pressure (>160/100 -may be rescreened)
* Estimated glomerular filtration rate (GFR)<30
* Malignancy (except squamous or basal cell of the skin) in the past 5 years
* MI, stroke or cardiovascular procedure within 12 months
* Known HIV positive or use of anti-HIV therapy (HAART)
* Unstable angina
* Significant pulmonary disease with oxygen dependency
* Chronic use (including in the past 6 months) of medications likely to cause weight gain or prevent weight loss (e.g. corticosteroids, lithium)
* Use of prescription weight loss medication or over-the-counter orlistat in the past 6 months
* Other serious medical condition likely to hinder accurate measurement of weight, or for which weight loss is contraindicated, or which would cause weight loss
* History of severe depression requiring hospitalization in the past 12 months
* Severe mental illness including bipolar disorder, schizophrenia or other psychotic disorders
* Current bulimia nervosa
* Unable or unwilling to use meal replacement products
* Consumption of >14 alcoholic drinks/week or > 5 drinks on more than 2 occasions in the past 12 months
* Use of illicit substances in the past 12 months
* Cigarette or cigar smoking in the past 2 months
* Pregnant or nursing within past 6 months
* Plans to become pregnant within 2 years
* Plans to relocate from the area within 1 year
* Another member of household is a study participant or staff in the trial

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to final data collection | Average time 6 months
  Participants will be followed until they reach 10% weight loss, anticipated average time 6 months, or up to 9 months.

SECONDARY OUTCOMES:
Change in insulin secretion | Average time 6 months
  Participants will be followed until they reach 10% weight loss, and anticipated average of 6 months, or up to 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M. Clark, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Result] Varma S, Lee CJ, Brown TT, Maruthur NM, Schweitzer M, Magnuson T, Kamel I, Clark JM. Comparative Effects of Medical Versus Surgical Weight Loss on Body Composition: a Pilot Randomized Trial. Obes Surg. 2019 Aug;29(8):2503-2510. doi: 10.1007/s11695-019-03879-4. PMID 30997619
- [Result] Lee CJ, Florea L, Sears CL, Maruthur N, Potter JJ, Schweitzer M, Magnuson T, Clark JM. Changes in Gut Microbiome after Bariatric Surgery Versus Medical Weight Loss in a Pilot Randomized Trial. Obes Surg. 2019 Oct;29(10):3239-3245. doi: 10.1007/s11695-019-03976-4. PMID 31256356